CLINICAL TRIAL: NCT03259308
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Parallel-group Efficacy and Safety Study of SHP647 as Induction Therapy in Subjects With Moderate to Severe Ulcerative Colitis (FIGARO UC 302)
Brief Title: Efficacy and Safety Study of SHP647 as Induction Therapy in Participants With Moderate to Severe Ulcerative Colitis
Acronym: FIGARO UC 302
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to discontinue the SHP647 (ontamalimab) clinical trial development program for inflammatory bowel diseases (IBD) early.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP647-302; 2017-000572-28 (EudraCT Number)
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Results first posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ontamalimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ontamalimab 25 mg (Experimental): Participants will receive 25 milligram (mg) of ontamalimab subcutaneous (SC) injection using a prefilled syringe (PFS) on Week 0, Week 4 and Week 8.
  Interventions: Drug: Ontamalimab
- Ontamalimab 75 mg (Experimental): Participants will receive 75 mg of ontamalimab SC injection using PFS on Week 0, Week 4 and Week 8.
  Interventions: Drug: Ontamalimab
- Placebo (Placebo Comparator): Participants will receive placebo matched to ontamalimab SC injection using PFS on Week 0, Week 4, and Week 8.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ontamalimab — Participants will receive 1 mL of ontamalimab sterile aqueous buffered solution at an appropriate concentration to provide the intended dose of drug (25 or 75 mg).
  Other Names: SHP647; PF- 00547659
  Arms: Ontamalimab 25 mg; Ontamalimab 75 mg
Drug: Placebo — Participants will receive 1 mL of sterile aqueous buffered solution.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of SHP647 in inducing remission, based on composite score of patient-reported symptoms and centrally read endoscopy, in participants with moderate to severe ulcerative colitis (UC).

DETAILED DESCRIPTION:
27Mar2020: Enrollment of new patients into this study has been paused due to the COVID-19 situation. The duration of this pause is dependent on the leveling and control of the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

- Participants and/or their parent or legally authorized representative must have an understanding, ability, and willingness to fully comply with study procedures and restrictions.

* Participants must be able to voluntarily provide written, signed, and dated informed consent and/or assent, as applicable, to participate in the study.
* Participants less than (<) 18 years of age must weigh >=40 kg and must have body mass index (BMI) >=16.5 kilogram per square metre (kg/m^2).
* Participants must have a documented diagnosis of UC for >=3 months before screening. The following must be available in each participant's source documentation:

  a. A biopsy report to confirm the histological diagnosis. b. A report documenting disease duration based upon prior colonoscopy. Note: If this documentation is not available at the time of screening, a colonoscopy with biopsy to confirm the diagnosis is required during the screening period.
* Participants must be willing to undergo a flexible sigmoidoscopy or colonoscopy, including biopsy sample collection, during screening after all other inclusion criteria have been met.
* Participants must have moderate to severe active UC, defined as a total Mayo score of >=6, including a centrally read endoscopic subscore >=2, rectal bleeding subscore >=1, and stool frequency subscore >=1 at baseline.
* Participants must have evidence of UC extending proximal to the rectum (ie, not limited to proctitis).
* Participants must have had an inadequate response to, or lost response to, or had an intolerance to at least 1 conventional treatment such as mesalamine (5-aminosalicylate [ASA]), glucocorticoids, immunosuppressants (azathioprine [AZA], 6-mercaptopurine [6-MP], or methotrexate [MTX]), or anti-tumor necrosis factor (TNF).
* Participants receiving any treatment(s) for UC are eligible provided they have been, and are anticipated to be, on a stable dose for the designated period of time.
* Participants are males or nonpregnant, nonlactating females who, if sexually active, agree to comply with the contraceptive requirements of the protocol, or females of nonchildbearing potential.

Exclusion Criteria:

* Participants with indeterminate colitis, microscopic colitis, non-steroidal anti-inflammatory drug-induced colitis, ischemic colitis, infectious colitis, or clinical/histologic findings suggestive of Crohn's disease.
* Participants with colonic dysplasia or neoplasia. (Participants with prior history of adenomatous polyps will be eligible if the polyps have been completely removed.)
* Participants with past medical history or presence of toxic megacolon.
* Participants with colonic stricture, past medical history of colonic resection, a history of bowel surgery within 6 months before screening, or who are likely to require surgery for UC during the treatment period.
* Participants at risk for colorectal cancer must have a colonoscopy performed during the screening period with results available within 10 days before the baseline visit, unless the participant has had a surveillance colonoscopy performed within 1 year prior to screening, and any adenomatous polyps found at that examination have been excised. Colonoscopy report and pathology report (if biopsies are obtained) from the colonoscopy performed during screening or in the prior year confirming no evidence of dysplasia and colon cancer must be available in the source documents.

Participants at risk for colorectal cancer include, but are not limited to:

1. Participants with extensive colitis for >=8 years or disease limited to left side of colon (ie, distal to splenic flexure) for >=10 years before screening, regardless of age.
2. Participants >=50 years of age at the time of signing of the informed consent form.

   - Participants have had prior treatment with ontamalimab (formerly PF-00547659, SHP647).

   - Participants with known or suspected intolerance or hypersensitivity to the investigational product(s), closely related compounds, or any of the stated ingredients.

   - Participants have received anti-TNF treatment within 60 days before baseline.

   - Participants have received any biologic with immunomodulatory properties (other than anti-TNFs) within 90 days before baseline.

   - Participants have received any nonbiologic treatment with immunomodulatory properties (other than their current background UC treatment) within 30 days before baseline.

   - Participants have ever received anti-integrin/adhesion molecule treatment (example (eg): natalizumab, vedolizumab, efalizumab, etrolizumab, or any other investigational anti-integrin/adhesion molecule).
   * Participants have received parenteral or rectal glucocorticoids, or rectal 5-ASA, within 14 days before screening endoscopic procedure.
   * Participants have received leukocyte apheresis or selective lymphocyte, monocyte, or granulocyte apheresis or plasma exchange within 30 days before baseline.
   * Participants have participated in other investigational studies within either 30 days or 5 half-lives of investigational product used in the study (whichever is longer) before baseline.
   * Participants have received a live (attenuated) vaccine within 30 days before the baseline visit.
   * Participants with active enteric infections (positive stool culture and sensitivity), Clostridium difficile infection or pseudomembranous colitis [Participants with C. difficile infection at screening may be allowed re-test after treatment], evidence of active cytomegalovirus infection or Listeria monocytogenes, known active invasive fungal infections such as histoplasmosis or parasitic infections, clinically significant underlying disease that could predispose the participants to infections, or a history of serious infection (requiring parenteral antibiotic and/or hospitalization) within 4 weeks before the baseline visit.
   * Participants with abnormal chest x-ray findings at screening, such as presence of active tuberculosis (TB), general infections, heart failure, or malignancy.
   * Participants with evidence of active or latent infection with Mycobacterium TB or participants with this history who have not completed a generally accepted full course of treatment before randomization are excluded. All other participants must have either the Mantoux (purified protein derivative [PPD]) tuberculin skin test or interferon gamma release assay (IGRA) performed.

Participants who have no history of previously diagnosed active or latent TB are excluded if they have a positive Mantoux (PPD) tuberculin skin test (ie >=5 millimeter [mm] induration) or a positive IGRA (the latter to be tested at the site's local laboratory) during screening or within 12 weeks before screening. If IGRA test cannot be performed locally, a central laboratory may be used, with prior agreement from the sponsor.

1. An IGRA is strongly recommended for participants with a prior Bacillus Calmette-Guerin (BCG) vaccination, but may be used for any participant. Documentation of IGRA product used and the test result must be in the participant's source documentation if performed locally. Acceptable IGRA products include QuantiFERON TB Gold Plus In-Tube Test.
2. If the results of the IGRA are indeterminate, the test may be repeated, and if a negative result is obtained, enrollment may proceed. In participants with no history of treated active or latent TB, a positive test on repeat will exclude the participant. Participants with a history of active or latent TB infection must follow instructions for "Participants with a prior diagnosis of active or latent TB are excluded unless both of the following criteria are met" in this criterion.
3. Participants with repeat indeterminate IGRA results, with no prior TB history, may be enrolled after consultation with a pulmonary or infectious disease specialist who determines low risk of infection (ie, participant would be acceptable for immunosuppressant [eg, anti-TNF] treatment without additional action). This consultation must be included in source documentation.

Results from a chest x-ray, taken within the 12 weeks before or during screening must show no abnormalities suggestive of active TB infection as determined by a qualified medical specialist.

Participants with a prior diagnosis of active or latent TB are excluded unless both of the following criteria are met:

1. The participant has previously received an adequate course of treatment for either latent (eg, 9 months of isoniazid or an acceptable alternative regimen, in a locale where rates of primary multidrug TB resistance are <5%. Participants from regions with higher rates of primary multidrug TB resistance are excluded) or active (acceptable multidrug regimen) TB infection. Evidence of diagnosis and treatment must be included in source documentation. Consultation with a pulmonary or infectious disease specialist to confirm adequate treatment (ie, participant would be acceptable for immunosuppressant [eg, anti-TNF] treatment without additional action) must be performed during the screening period. The consultation report must be included in source documentation prior to enrollment.
2. A chest x-ray performed within 12 weeks before screening or during screening indicates no evidence of active or recurrent disease, and documentation of interpretation by a qualified medical specialist must be included in source documentation.

   * Participants with a pre-existing demyelinating disorder such as multiple sclerosis or new onset seizures, unexplained sensory motor, or cognitive behavioral, neurological deficits, or significant abnormalities noted during screening.
   * Participants with any unexplained symptoms suggestive of progressive multifocal leukoencephalopathy (PML) based on the targeted neurological assessment during the screening period.
   * Participants with a transplanted organ. Skin grafts to treat pyoderma gangrenosum are allowed.
   * Participants with a significant concurrent medical condition at the time of screening or baseline, including, but not limited to, the following:

<!-- -->

1. Any major illness/condition or evidence of an unstable clinical condition (eg, renal, hepatic, hematologic, gastrointestinal (except disease under study), endocrine, cardiovascular, pulmonary, immunologic [eg, Felty's syndrome], or local active infection/infectious illness) that, in the investigator's judgment will substantially increase the risk to the participant if he or she participates in the study.
2. Cancer or history of cancer or lymphoproliferative disease within the previous 5 years (other than resected cutaneous basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the uterine cervix that has been treated with no evidence of recurrence).
3. Presence of acute coronary syndrome (eg, acute myocardial infarction, unstable angina pectoris) within 24 weeks before screening.
4. History of significant cerebrovascular disease within 24 weeks before screening.

   - Participants who have had significant trauma or major surgery within 4 weeks before the screening visit, or with any major elective surgery scheduled to occur during the study.

   - Participants with evidence of cirrhosis with or without decompensation.

   - Participants with primary sclerosing cholangitis.

   - Participants with evidence of positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb).

   Note: If a participant tests negative for HBsAg, but positive for HBcAb, the participant would be considered eligible if no presence of hepatitis B virus (HBV) DNA is confirmed by HBV DNA polymerase chain reaction (PCR) reflex testing performed in the central laboratory.
   * Participants with chronic hepatitis C virus (HCV) (positive HCV antibody [HCVAb] and HCVRNA).

   Note: Participants who are HCVAb positive without evidence of HCV RNA may be considered eligible (spontaneous viral clearance or previously treated and cured [defined as no evidence of HCVRNA at least 12 weeks prior to baseline]).
   * Participants with any of the following abnormalities in hematology and/or serum chemistry profiles during screening.

   Note: Screening laboratory tests, if the results are considered by the investigator to be transient and inconsistent with the participant's clinical condition, may be repeated once during the screening period for confirmation. Results must be reviewed for eligibility prior to the screening endoscopy procedure.

<!-- -->

1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels >=3.0×upper limit of normal (ULN).
2. Total bilirubin level >=1.5×ULN or >2.0×ULN if the participant has a known documented history of Gilbert's syndrome.
3. Hemoglobin level <=80 gram per liter (g/L) (8.0 gram per deciliter [g/dL]).
4. Platelet count <=100×10^9 per liter (/L) (100,000 cells per cubic millimeter [mm^3]) or >=1000×10^9/L (1,000,000 cells/mm^3).
5. White blood cell count <=3.5×10^9/L (3500 cells/mm^3).

   - Absolute neutrophil count (ANC)<2×10^9/L (2000 cells/mm^3).

   - Serum creatinine level >1.5 × ULN or estimated glomerular filtration rate <30 ml/min/1.73m^2 based on the abbreviated Modification of Diet in Renal Disease Study Equation.

   Note: If platelet count is <150,000 cells/mm^3, a further evaluation should be performed to rule out cirrhosis, unless another etiology has already been identified.
   * Participants with known human immunodeficiency virus (HIV) infection based on documented history, with positive serological test, or positive HIV serologic test at screening, tested at the site's local laboratory in accordance with country requirements or tested at the central laboratory.

   Note: A documented negative HIV test within 6 months of screening is acceptable and does not need to be repeated.

   - Participants who have, or who have a history of (within 2 years before screening), serious psychiatric disease, alcohol dependency, or substance/drug abuse or dependency of any kind, including abuse of medical marijuana (cannabis).

   - Participants with any other severe acute or chronic medical or psychiatric condition or laboratory or electrocardiogram (ECG) abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

   - Female participants who are planning to become pregnant during the study period.
   * Participants who do not agree to postpone donation of any organ or tissue, including male participants who are planning to bank or donate sperm and female participants who are planning to harvest or donate eggs, for the duration of the study and through 16 weeks after last dose of investigational product.
   * Participants who are investigational site staff members or relatives of those site staff members or Participants who are Shire employees directly involved in the conduct of the study.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (207):
- United States (62):
  - Arizona Digestive Health Mesa - East, Mesa, Arizona
  - Elite Clinical Studies - Phoenix - Clinedge - PPDS, Phoenix, Arizona
  - Advanced Research Center, Anaheim, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - United Medical Doctors, Encinitas, California
  - University of California San Diego, La Jolla, California
  - VA Long Beach Healthcare System - NAVREF - PPDS, Long Beach, California
  - Facey Medical Foundation, Mission Hills, California
  - United Medical Doctors, Murrieta, California
  - Alliance Clinical Research-(Vestavia Hills), Poway, California
  - University of California San Francisco, San Francisco, California
  - Care Access Research, San Pablo, San Pablo, California
  - Renaissance Research Medical Group, INC, Cape Coral, Florida
  - Gastro Florida, Clearwater, Florida
  - Hi Tech and Global Research, LLc, Coral Gables, Florida
  - ENCORE Borland-Groover Clinical Research - ERN - PPDS, Jacksonville, Florida
  - SIH Research, Kissimmee, Florida
  - Alliance Medical Research LLC, Lighthouse PT, Florida
  - Sanchez Clinical Research, Inc, Miami, Florida
  - Crystal Biomedical Research, Miami Lakes, Florida
  - Pharma Research International Inc, Naples, Florida
  - Bayside Clinical Research - New Port Richey, New Port Richey, Florida
  - Accel Research Sites - St. Petersburg - ERN - PPDS, Pinellas Park, Florida
  - BRCR Medical Center Inc., Plantation, Florida
  - DBC Research, Tamarac, Florida
  - Infinite Clinical Trials, Atlanta, Georgia
  - Atlanta Center For Gastroenterology PC, Decatur, Georgia
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Loretto Hospital, Chicago, Illinois
  - IL Gastroenterology Group, Gurnee, Illinois
  - Edward Hines Jr VA Hospital - NAVREF - PPDS, Hines, Illinois
  - Dupage Medical Group, Oakbrook Terrace, Illinois
  - Gastroenterology Associates of Hazard, Hazard, Kentucky
  - CroNOLA, LLC., Houma, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Commonwealth Clinical Studies LLC, Brockton, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - National Clinical, LLC, Hamtramck, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - St Louis Center For Clinical Research, St Louis, Missouri
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Encompass Care, North Las Vegas, Nevada
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - Weill Cornell Medical College, New York, New York
  - Southtowns Gastroenterology, PLLC, Orchard Park, New York
  - East Carolina Gastroenterology, Jacksonville, North Carolina
  - Prestige Clinical Research, Franklin, Ohio
  - Ohio Clinical Research Partners LLC, Mentor, Ohio
  - Veteran's Research and Education Foundation - NAVREF - PPDS, Oklahoma City, Oklahoma
  - Veterans Research Foundation of Pittsburgh - NAVREF - PPDS, Pittsburgh, Pennsylvania
  - Digestive Health Associates of Texas, P.A.dba DHAT Research Institute, Garland, Texas
  - Precision Research Institute, LLC, Houston, Texas
  - Biopharma Informatic Inc., Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Aztec Medical Research, Houston, Texas
  - BI Research Center, Houston, Texas
  - Southern Star Research Institute LLC, San Antonio, Texas
  - Mid Atlantic Health Specialists, Galax, Virginia
  - Winchester Gastroenterology Associates, Winchester, Virginia
  - Mayo Clinic Health System - PPDS, La Crosse, Wisconsin
- Argentina (3):
  - Sanatorio 9 de Julio SA, San Miguel de Tucumán, Tucumán Province
  - Fundación Favaloro, Buenos Aires
  - Hospital Privado Centro Médico de Córdoba, Córdoba
- Belgium (4):
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Gasthuisberg, Leuven, Vlaams Brabant
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - CHU Mouscron, Mouscron
- Clinical Center Banja Luka, Banja Luka, Bosnia and Herzegovina
- Bulgaria (13):
  - Second Multiprofile Hospital for Active Treatment Sofia, Sofia, Sofia-Grad
  - Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia, Sofia-Grad
  - University Multiprofile Hospital for Active Treatment Sveta Anna, Sofia, Sofia-Grad
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment EOOD, Sofia, Sofia-Grad
  - University Multiprofile Hospital for Active Treatment - Dr. Georgi Stranski EAD, Pleven
  - Multiprofile Hospital for Active Treatment Eurohospital, Plovdiv
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases Dr.D.Gramatikov- Ruse- PPDS, Rousse
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - Medical Center Excelsior OOD - PPDS, Sofia
  - University Multiprofile Hospital for Active Treatment Sv Ivan Rilski EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - Medical Center Convex EOOD, Sofia
  - Diagnostic Consultative Centre Mladost - M OOD, Varna
- Canada (2):
  - Percuro Clinical Research LTD, Victoria, British Columbia
  - Toronto Digestive Disease Associates Inc, Toronto, Ontario
- Colombia (4):
  - Hospital Pablo Tobón Uribe, Medellín, Antioquia
  - Fundación Clínica Shaio, Bogota, Cundinamarca
  - Servimed S.A.S, Bucaramanga, Santander Department
  - IPS Centro Médico Julián Coronel S.A.S. - PPDS, Cali
- Estonia (3):
  - East Viru Central Hospital, Kohta-Järve
  - OÜ LV Venter, Pärnu
  - West Tallinn Central Hospital, Tallinn
- Greece (4):
  - Ippokrateio General Hospital of Athens, Athens, Attica
  - University General Hospital of Patras, Pátrai
  - Theageneio Anticancer Oncology Hospital of Thessaloniki, Thessaloniki
  - Euromedica - PPDS, Thessaloniki
- Hungary (12):
  - Bekes Megyei Kozponti Korhaz, Békéscsaba
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Pannónia Magánorvosi Centrum Kft, Budapest
  - ENDOMEDIX Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bekes Megyei Kozponti Korhaz, Gyula
  - Mohacsi Korhaz, Mohács
  - Tolna Megyei Balassa János Kórház, Szekszárd
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz, Szentes
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Jávorszky Ödön Kórház, Vác
  - Csolnoky Ferenc Korhaz, Veszprém
- St Vincent's University Hospital, Dublin, Ireland
- Japan (17):
  - Sapporo Medical University Hospital, Sapporo, Hokkaidô
  - Medical Corporation Aoyama Clinic, Kobe, Hyôgo
  - Hyogo College of Medicine, Nishinomiya-shi, Hyôgo
  - Kunimoto Hospital, Asahikawa
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Aizawa Hospital, Matsumoto-shi
  - Chiinkai Dojima General & Gastroenterology Clinic, Osaka
  - Kinshukai Infusion Clinic, Osaka
  - Yodogawa Christian Hospital, Osaka
  - Ishida Clinic of IBD and Gastroenterology, Ōita
  - Bellland General Hospital, Sakai
  - Toho University Sakura Medical Center, Sakura
  - Tohoku Rosai Hospital, Sendai
  - Dokkyo Medical University Hospital, Shimotsuga-gun
  - Medical Corporation Shoyu-kai Fujita Gastroenterology Hospital, Takatsuki
  - Nihonbashi Egawa Clinic, Tokyo
  - Koukokukai Ebisu Clinic, Tokyo
- Lebanon (2):
  - Rafik Hariri University Hospital, Beirut
  - Hammoud Hospital University Medical Center, Saida
- Mexico (11):
  - Health Pharma Professional Research S.A de C.V., Mexico City, Mexico City
  - Clinica de Higado y Gastroenterologia Integral, S.C., Cuernavaca, Morelos
  - JM Research S.C, Cuernavaca, Morelos
  - Unidad de Atencion Medica e Investigacion en Salud, Mérida, Yucatán
  - Centro de Investigación Médica Aguascalientes, Aguascalientes
  - Phylasis Clinicas Research S. de R.L. de C.V., Cuautitlán Izcalli
  - Centro de Investigacion Clinica Acelerada, S.C., Distrito Federal
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Accelerium, S. de R.L. de C.V., Monterrey
  - Clinical Research Institute, Tlalnepantla
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Zapopan, Jalisco
- New Zealand (4):
  - Auckland City Hospital, Grafton, Auckland
  - Dunedin Hospital, Dunedin, South Island
  - Wellington Hospital, Newtown, Wellington Region
  - Waikato Hospital, Hamilton
- Portugal (5):
  - Hospital de Braga, Braga
  - Hospital Senhora da Oliveira - Guimaraes, E.P.E, Guimarães
  - Hospital da Luz, Lisbon
  - Centro Hospitalar do Algarve - Hospital de Portimao, Portimão
  - Hospital de São Bernardo, Setúbal
- Slovakia (3):
  - Univerzitna nemocnica Bratislava, Bratislava
  - KM Management, spol. s r.o., Nitra
  - Gastro LM, s.r.o., Prešov
- South Korea (16):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gang'weondo
  - CHA Bundang Medical Center, CHA University, Seongnam, Gyeonggido
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggido
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center PPDS, Seoul
  - Inje University Seoul Paik Hospital, Seoul
- Spain (10):
  - C.H. Regional Reina Sofia - PPDS, Córdoba, Córdoba
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Centro Medico Teknon - Grupo Quironsalud, Barcelona
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Universität Zürich, Zurich, Zürich (de), Switzerland
- Turkey (Türkiye) (2):
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Mersin University Medical Faculty, Mersin
- Ukraine (27):
  - Regional Municipal Non-profit Enterprise "Chernivtsi Regional Clinical Hospital", Chernivtsi, Chernivtsi Oblast
  - Municipal Nonprofit Enterprise CCH #2 n.a. prof. O.O. Shalimov of Kharkiv City Council, Kharkiv, Kharkivs’ka Oblast’
  - Municipal Nonprofit Enterprise Vinnytsia City Clinical Hospital #1, Vinnytsia, Vinnytsia Oblast
  - Communal Nonprofit Enterprise Vinnytsia Regional Clinical Hospital named after N.I. Pirogov VRC, Vinnytsia, Vinnytsia Oblast
  - ME Dnipropetrovsk Regional Clinical Hospital n.a. I.I Mechnykov Dnipropetrovsk Regional Council, Dnipro
  - LLC Medical Center Family Medicine Clinic, Dnipro
  - State Institution "Institute of Gastroenterology of National Academy of Medical Sciences of Ukraine", Dnipro
  - Clinic of SI National Institute of Therapy n.a. L.T. Mala of NAMS of Ukraine, Kharkiv
  - Communal Non-Commercial Enterprize of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - MNPE of Kharkiv Regional Council Regional Clinical Specialized Dispensary of Radiation Protection, Kharkiv
  - Municipal Non-profit Enterprise Kherson City Clinical Hospital named after Ye.Ye. Karabelesh, Kherson
  - Municipal Enterprise Kryvyi Rih City Clinical Hospital #2 of Kryvyi Rih City Council, Kryvyi Rih
  - Medical Center of LLC Medical Clinic Blagomed, Kyiv
  - Kyiv City Clinical Hospital #18, Kyiv
  - Treatment and Diagnostic Center "Healthy and Happy" of LLC "Healthy and Happy", Kyiv
  - Municipal Institution of KRC Kyiv Regional Hospital #2, Kyiv
  - Municipal Non-profit Enterprise of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv
  - Lviv Railway Clinical Hospital of branch Health Center of Joint Stock Co. Ukrainian Railway, Lviv
  - Municipal Nonprofit Enterprise Lviv Clinical Emergency Care Hospital, Lviv
  - Municipal Non-profit Enterprise Odessa Regional Clinical Hospital of Odessa Regional Council, Odesa
  - MNPE Central City Clinical Hospital of Uzhhorod City Council, Uzhhorod
  - Medical Clinical Research Center of Medical Center LLC Health Clinic, Vinnytsia
  - Communal Nonprofit Enterprise Vinnytsia Regional Clinical Hospital named after N.I. Pirogov VRC, Vinnytsia
  - City Clinical Hospital #1, Vinnytsia
  - Communal Non-Commercial Enterprise "Vinnytsia City Clinical Hospital №1", Vinnytsia
  - Municipal Non-profit Enterprise City Emergency Care Hospital of Zaporizhzhia Regional Council, Zaporizhzhia
  - MNPE City Hospital No. 6 of Zaporizhzhia City Council, Zaporizhzhia

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fde4db2bf003ab4741c

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 205 sites between 5 December 2017 (first participant first visit) and 06 October 2020 (last participant last visit).
Pre-assignment Details: A total of 279 participants were enrolled and randomized in this study.
Groups:
- Placebo: Participants received placebo matched to ontamalimab subcutaneous (SC) injection, using a prefilled syringe (PFS) on Week 0, Week 4, and Week 8 in a 12-week treatment period.
- Ontamalimab 25 mg: Participants received 25 milligrams (mg) of ontamalimab SC injection, using a PFS on Week 0, Week 4 and Week 8 in a 12-week treatment period.
- Ontamalimab 75 mg: Participants received 75 mg of ontamalimab SC injection, using a PFS on Week 0, Week 4 and Week 8 in a 12-week treatment period.
Period: Overall Study
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Started | 56 | 111 | 112
Completed | 49 | 103 | 105
Not Completed | 7 | 8 | 7
Not completed — Adverse Event | 5 | 4 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Protocol Deviation | 0 | 3 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety set consisted of all participants who had received at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg | Total
Number analyzed (Participants) | 56 | 111 | 112 | 279
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.6 (13.50) | 43.5 (14.16) | 43.9 (13.08) | 43.3 (13.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 46 | 45 | 114
  Male | 33 | 65 | 67 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 17 | 16 | 38
  Not Hispanic or Latino | 51 | 93 | 96 | 240
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 5 | 3 | 8
  Race: Asian: Japanese | 6 | 5 | 6 | 17
  Race: Asian: Korean | 4 | 5 | 8 | 17
  Race: Asian: Other | 1 | 0 | 0 | 1
  Race: Black or African American | 2 | 4 | 1 | 7
  Race: White | 41 | 85 | 88 | 214
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Race: Multiple | 1 | 5 | 1 | 7
  Race: Other (Unspecified) | 1 | 1 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Remission Based on Composite Score at Week 12
Description: Remission was defined as a composite score of patient-reported symptoms using daily e-diary and centrally read endoscopy as stool frequency sub-score of 0 or 1 with at least a 1-point change from baseline, rectal bleeding sub-score of 0 and endoscopic sub-score of 0 or 1 (modified, excluded friability). The composite score was a recommended measure derived from the Mayo score without the physician global assessment (PGA) sub-score and ranged from 0 to 9 points. The Mayo score was a measure of Ulcerative Colitis (UC) disease activity. It ranged from 0 to 12 points and consisted of 4 sub-scores, each graded from 0 to 3 with higher scores indicating more severe disease. The sub-scores were stool frequency (0-3); rectal bleeding (0-3); findings of endoscopy (0-3); PGA (0-3).
Time Frame: At Week 12
Population: Full analysis set (FAS) consisted of all participants in the randomized set who had received at least 1 dose of investigational product (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 56 | 111 | 112
Participants | 7 | 30 | 33
Statistical Analysis 1: Comparison: Placebo vs Ontamalimab 25 mg; Test type: Superiority; p = 0.027, Cochran-Mantel-Haenszel; P-value was based on Cochran-Mantel-Haenszel chi-square test stratified by actual status of prior anti-TNF treatment and glucocorticoid at baseline
Statistical Analysis 2: Comparison: Placebo vs Ontamalimab 75 mg; Test type: Superiority; p = 0.014, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With Endoscopic Remission at Week 12
Description: Endoscopic remission was defined by centrally read endoscopic sub-score 0 or 1 (modified, excluded friability). The centrally read endoscopic sub-score of Mayo score ranged from 0 to 3 with higher scores indicating more severe disease.
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 56 | 111 | 112
Participants | 7 | 39 | 38
Statistical Analysis 1: Comparison: Placebo vs Ontamalimab 25 mg; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ontamalimab 75 mg; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With Clinical Remission at Week 12
Description: Clinical remission was defined by stool frequency sub-score of 0 or 1 with at least a 1-point change from baseline in stool frequency sub-score, and rectal bleeding sub-score of 0. The stool frequency sub-score and rectal bleeding sub-score ranged from 0 to 3 with higher scores indicating more severe disease.
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 56 | 111 | 112
Participants | 10 | 50 | 56
Statistical Analysis 1: Comparison: Placebo vs Ontamalimab 25 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ontamalimab 75 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Clinical Response Based on Composite Score at Week 12
Description: Clinical response based on composite score was defined as a decrease from baseline in the composite score of patient-reported symptoms using daily e-diary and centrally read endoscopy of at least 2 points and at least 30 percent (%), with an accompanying decrease in the sub-score for rectal bleeding greater than or equal to (>=) 1 point or a sub-score for rectal bleeding less than or equal to (<=) 1. The composite score was a recommended measure derived from the Mayo score without the PGA sub-score and ranged from 0 to 9 points. The Mayo score was a measure of UC disease activity. It ranged from 0 to 12 points and consisted of 4 sub-scores, each graded from 0 to 3 with higher scores indicating more severe disease The sub-scores were stool frequency (0-3); rectal bleeding (0-3); findings of endoscopy (0-3); PGA (0-3).
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 56 | 111 | 112
Participants | 16 | 67 | 64
Statistical Analysis 1: Comparison: Placebo vs Ontamalimab 25 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ontamalimab 75 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With Mucosal Healing Based on Endoscopic and Histological Assessment Using the Geboes Score Grading System at Week 12
Description: Mucosal healing was defined by centrally read endoscopic sub-score 0 or 1 (modified, excluded friability) and centrally read Geboes score of <=2. The centrally read endoscopic sub-score of Mayo score ranged from 0 to 3 with higher scores indicating more severe disease. Geboes score grading system, was a validated score for evaluating histologic disease activity in UC as follows: grade 0 equal to (=) structural and architectural changes; grade 1 = chronic inflammatory infiltrate; grade 2 = lamina propria neutrophils and eosinophils; grade 3 = neutrophils in the epithelium; grade 4 = crypt destruction; grade 5 = erosions or ulceration. A higher Geboes score indicating more severe disease. Number of participants with mucosal healing based on endoscopic and histological assessment using the Geboes score grading system were reported.
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 56 | 111 | 112
Participants | 6 | 35 | 30
Statistical Analysis 1: Comparison: Placebo vs Ontamalimab 25 mg; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Ontamalimab 75 mg; Test type: Superiority; p = 0.017, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants With Remission Based on Total Mayo Score at Week 12
Description: Remission was defined as a Total Mayo score of <=2 with no individual sub-score (stool frequency, rectal bleeding, endoscopy [modified, excluded friability], and PGA) exceeding 1, at the Week 12. The Total Mayo score ranged from 0 to 12 points and consisted of 4 sub-scores, each graded from 0 to 3 with higher scores indicating more severe disease: stool frequency (0-3); rectal bleeding (0-3); findings of endoscopy (0-3); PGA (0-3).
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 56 | 111 | 112
Participants | 5 | 28 | 26

7. Secondary Outcome: Number of Participants With Clinical Response Based on Total Mayo Score at Week 12
Description: Clinical response (Mayo) was defined as a decrease from baseline in the Total Mayo score of at least 3 points and at least 30%, with an accompanying decrease in the sub-score for rectal bleeding >=1 point or an absolute sub-score for rectal bleeding <=1. The Total Mayo score ranged from 0 to 12 points and consisted of the following 4 sub-scores, each graded from 0 to 3 with higher scores indicating more severe disease: stool frequency (0-3); rectal bleeding (0-3); findings of endoscopy (0-3); PGA (0-3).
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 56 | 111 | 112
Participants | 19 | 66 | 63

8. Secondary Outcome: Number of Participants With Partial Mayo Score <=2 With no Individual Sub-score Greater Than (>) 1 at Weeks 4, 8, and 12
Description: The partial Mayo score ranged from 0 to 9 points and consisted of the following 3 sub-scores, each graded from 0 to 3 with higher scores indicating more severe disease: Stool frequency (0-3); Rectal bleeding (0-3); PGA (0-3). The partial Mayo score did not include the endoscopy sub-score.
Time Frame: At Weeks 4, 8, and 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 56 | 111 | 112
Participants
  At Week 4 | 6 | 26 | 23
  At Week 8 | 12 | 53 | 41
  At Week 12 | 10 | 49 | 52

9. Secondary Outcome: Number of Participants With Clinical Remission With Stool Frequency Sub-scores of 0 or 1 and Rectal Bleeding Sub-score of 0 at Weeks 4 and 8
Description: Number of participants were reported with stool frequency sub-scores of 0 or 1 and rectal bleeding sub-score of 0. Clinical remission was defined as stool frequency sub-score of 0 or 1 with at least a 1-point change from baseline in stool frequency sub-score, and a rectal bleeding sub-score of 0. The stool frequency sub-score and rectal bleeding sub-score of Mayo score ranges from 0 to 3 with higher scores indicating more severe disease.
Time Frame: At Weeks 4 and 8
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 56 | 111 | 112
Participants
  At Week 4 | 4 | 28 | 22
  At Week 8 | 10 | 52 | 56

10. Secondary Outcome: Number of Participants With Endoscopic Remission With Sub-score of 0 at Week 12
Description: Endoscopic remission was defined by centrally read endoscopic sub-score 0 (modified, excluded friability). The centrally read endoscopic sub-score of Mayo score ranged from 0 to 3 with higher scores indicating more severe disease.
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 56 | 111 | 112
Participants | 1 | 14 | 14

11. Secondary Outcome: Number of Participants With Clinical Remission With Both Rectal Bleeding and Stool Frequency Sub-scores of 0 at Weeks 4, 8, and 12
Description: Number of participants were reported with rectal bleeding and stool frequency sub-scores of 0. Clinical remission was defined as both rectal bleeding and stool frequency sub-scores of 0. The stool frequency sub-score and rectal bleeding sub-score of Mayo score ranges from 0 to 3 with higher scores indicating more severe disease.
Time Frame: At Weeks 4, 8, and 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 56 | 111 | 112
Participants
  At Week 4 | 0 | 15 | 12
  At Week 8 | 5 | 29 | 19
  At Week 12 | 6 | 36 | 26

12. Secondary Outcome: Number of Participants With Deep Remission at Week 12
Description: Deep remission was defined as both endoscopic and rectal bleeding sub-scores of 0, and stool frequency sub-score <=1 and a centrally read Geboes score of <=2. The stool frequency sub-score, rectal bleeding sub-score and endoscopic sub-score of Mayo score ranged from 0 to 3 with higher scores indicating more severe disease. The composite score was a recommended measure consisted of the Mayo score without the PGA sub-score and ranged from 0 to 9 points. Geboes score grading system was a validated score for evaluating histologic disease activity in UC as follows: grade 0 = structural and architectural changes; grade 1 = chronic inflammatory infiltrate; grade 2 = lamina propria neutrophils and eosinophils; grade 3 = neutrophils in the epithelium; grade 4 = crypt destruction; grade 5 = erosions or ulceration. A higher Geboes score indicating more severe disease.
Time Frame: At Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 56 | 111 | 112
Participants | 1 | 11 | 9

13. Secondary Outcome: Change From Baseline in Average Worst Abdominal Pain Score Based on Patient Reported Outcome-ulcerative Colitis (PRO-UC) Daily e-Diary at Week 12
Description: PRO-UC signs and symptom data were collected using a daily e-diary during treatment period. Collection of daily e-diary data was begun at least 10 days before the baseline visit. Participants were asked to record the signs and symptom data of abdominal pain worst severity, as experienced over the previous 24 hours, in the e-diary. Participant's signs and symptom average scores at each scheduled visit were calculated based on data recorded over the most recent 3 days (consecutive or non-consecutive) of last 10 days prior to the scheduled visit start date excluding the following days: day of any bowel preparation, day of endoscopy, any days between day of bowel preparation and day of endoscopy, and the 2 days after the day of endoscopy. Abdominal pain's worst severity assessment was based on an 11-point numerical rating scale with 0 anchor at "No pain" and 10 at "Worst Imaginable Pain" as experienced over the previous 24 hours, in the e-diary. Higher scores indicating more severe pain.
Time Frame: Baseline, Week 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 47 | 104 | 107
Score on a Scale | -1.69 (0.309) | -2.49 (0.218) | -1.83 (0.215)

14. Secondary Outcome: Change From Baseline in Diarrhea (Average Loose Bowel Movements) Score Based on PRO-UC Daily e-Diary at Week 12
Description: PRO-UC signs and symptom data were collected using a daily e-diary during treatment period. Collection of daily e-diary data was begun at least 10 days before the baseline visit. Participants were asked to record the signs and symptom data for number of loose bowel movement, as experienced over the previous 24 hours, in the e-diary. Participant's signs and symptom average scores at each scheduled visit were calculated based on data recorded over the most recent 3 days (consecutive or nonconsecutive) of the last 10 days prior to the scheduled visit start date excluding the following days: day of any bowel preparation, day of endoscopy, any days between day of bowel preparation and day of endoscopy, and the 2 days after the day of endoscopy. Average number of loose bowel movement ranged from 0-27. Higher scores indicating more frequent bowel movements.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 47 | 104 | 107
Score on a Scale | -1.41 (0.405) | -3.50 (0.286) | -2.87 (0.284)

15. Secondary Outcome: Change From Baseline in Average Bowel Movements With Urgency Score Based on PRO-UC Daily e-Diary at Week 12
Description: PRO-UC signs and symptom data were collected using a daily e-diary during treatment period. Collection of daily e-diary data was begun at least 10 days before the baseline visit. Participants were asked to record the signs and symptom data for number of bowel movement with urgency, as experienced over the previous 24 hours. Participant's signs and symptom average scores at each scheduled visit were calculated based on data recorded over the most recent 3 days (consecutive or nonconsecutive) of the last 10 days prior to the scheduled visit start date excluding the following days: day of any bowel preparation, day of endoscopy, any days between day of bowel preparation and day of endoscopy, and the 2 days after the day of endoscopy. Average number bowel movements urgency ranged from 0 to 27. Higher scores indicating more frequent bowel movements.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 47 | 104 | 107
Score on a Scale | -1.09 (0.373) | -2.87 (0.263) | -2.56 (0.264)

16. Secondary Outcome: Change From Baseline in Absolute Stool Frequency (Average Number of Bowel Movements) Score Based on PRO-UC Daily e-Diary at Week 12
Description: PRO-UC signs and symptom data were collected using a daily e-diary during treatment period. Collection of daily e-diary data was begun at least 10 days before the baseline visit. Participants were asked to record the signs and symptom data for average number of bowel movements, as experienced over the previous 24 hours. Participant's signs and symptom average scores at each scheduled visit were calculated based on data recorded over the most recent 3 days (consecutive or nonconsecutive) of the last 10 days prior to the scheduled visit start date excluding the following days: day of any bowel preparation, day of endoscopy, any days between day of bowel preparation and day of endoscopy, and the 2 days after the day of endoscopy. Average number bowel movements ranged from 0 to 27. Higher scores indicating more frequent bowel movements.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 47 | 104 | 107
Score on a Scale | -1.26 (0.386) | -3.32 (0.272) | -2.97 (0.272)

17. Secondary Outcome: Change From Baseline in Absolute Rectal Bleeding (Average Number Bowel Movements With Blood) Score Based on PRO-UC Daily e-Diary at Week 12
Description: PRO-UC signs and symptom data were collected using a daily e-diary during treatment period. Collection of daily e-diary data was begun at least 10 days before the baseline visit. Participants were asked to record the signs and symptom data for average number of bowel movements with blood, as experienced over the previous 24 hours. Participant's signs and symptom average scores at each scheduled visit were calculated based on data recorded over the most recent 3 days (consecutive or nonconsecutive) of the last 10 days prior to the scheduled visit start date excluding the following days: day of any bowel preparation, day of endoscopy, any days between day of bowel preparation and day of endoscopy, and the 2 days after the day of endoscopy. Average number bowel movements with blood ranged from 0 to 27. Higher scores indicating more frequent bowel movements with blood.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 47 | 104 | 107
Score on a Scale | -2.05 (0.379) | -3.74 (0.267) | -3.41 (0.265)

18. Secondary Outcome: Change From Baseline in Total Sign/Symptom Score Based on PRO-UC Daily e-Diary at Week 12
Description: Total sign/symptom score was the average of the average scores of worst abdominal pain over the past 24 hours and the conversion scale values for number of bowel movements blood, number of bowel movements with urgency, number of bowel movements and number of loose bowel movements, with scale ranged of 0-10, with higher scores indicating higher severity.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 47 | 104 | 107
Score on a Scale | -1.15 (0.246) | -2.32 (0.173) | -2.00 (0.172)

19. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Domains Scores at Weeks 8 and 12
Description: IBDQ was a psychometrically validated participant-reported outcome (PRO) instrument for measuring the disease-specific health-related quality of life (HRQL) in participants with inflammatory bowel disease, including UC. The IBDQ consisted of 32 items, which were grouped into 4 dimensions: bowel function, emotional status, systemic symptoms, and social function. The 4 domains were scored as follows: Bowel symptoms: 10 to 70; Systemic symptoms: 5 to 35; Emotional function: 12 to 84; Social function: 5 to 35. Higher scores indicating a better quality of life.
Time Frame: Baseline, Weeks 8 and 12
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure and number analyzed refer to participants evaluable at specific time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 53 | 108 | 106
Score on a Scale
  IBDQ Bowel Function Dimension Score: Change at Week 8 | 9.59 (1.611) | 16.66 (1.189) | 15.36 (1.180)
  IBDQ Bowel Function Dimension Score: Change at Week 12: number analyzed (Participants) | 50 | 104 | 106
  IBDQ Bowel Function Dimension Score: Change at Week 12 | 9.51 (1.707) | 17.71 (1.250) | 15.86 (1.232)
  IBDQ Emotional Status Dimension Score: Change at Week 8 | 8.91 (1.701) | 15.18 (1.255) | 14.41 (1.247)
  IBDQ Emotional Status Dimension Score: Change at Week 12: number analyzed (Participants) | 50 | 104 | 106
  IBDQ Emotional Status Dimension Score: Change at Week 12 | 9.94 (1.861) | 14.84 (1.359) | 14.73 (1.341)
  IBDQ Systemic Symptoms Dimension Score: Change at Week 8 | 3.84 (0.759) | 6.61 (0.561) | 5.86 (0.557)
  IBDQ Systemic Symptoms Dimension Score: Change at Week 12: number analyzed (Participants) | 50 | 104 | 106
  IBDQ Systemic Symptoms Dimension Score: Change at Week 12 | 3.85 (0.814) | 7.34 (0.596) | 6.04 (0.587)
  IBDQ Social Function Dimension Score: Change at Week 8 | 5.06 (0.873) | 6.97 (0.643) | 6.75 (0.640)
  IBDQ Social Function Dimension Score: Change at Week 12: number analyzed (Participants) | 50 | 104 | 106
  IBDQ Social Function Dimension Score: Change at Week 12 | 5.09 (0.926) | 7.68 (0.677) | 7.03 (0.668)

20. Secondary Outcome: Change From Baseline in IBDQ Total Scores at Weeks 8 and 12
Description: IBDQ was a psychometrically validated PRO instrument for measuring the disease-specific HRQL in participants with inflammatory bowel disease, included UC. The IBDQ consisted of 32 items, which were grouped into 4 dimensions: bowel function, emotional status, systemic symptoms, and social function. The 4 domains were scored as follows: Bowel symptoms: 10 to 70; Systemic symptoms: 5 to 35; Emotional function: 12 to 84; Social function: 5 to 35. The total IBDQ score ranged from 32 to 224. For the total score and each domain, a higher score indicating better HRQL. A score of at least 170 corresponds to clinical remission and an increase of at least 16 points was considered to indicate a clinically meaningful improvement.
Time Frame: Baseline, Weeks 8 and 12
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 53 | 108 | 106
Score on a Scale
  Change at Week 8 | 27.56 (4.574) | 45.63 (3.380) | 42.58 (3.358)
  Change at Week 12: number analyzed (Participants) | 50 | 104 | 106
  Change at Week 12 | 28.39 (4.990) | 47.75 (3.649) | 43.85 (3.604)

21. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF-36), Version 2, Acute (Physical and Mental Component Summary Scores) at Week 12
Description: SF-36 was a generic quality-of-life instrument that had been widely used to assess health-related quality of life (HRQL) of participants. SF-36 consisted of 36 items that were aggregated into 8 multi-item scales (physical functioning [1=yes, limited a lot to 3=no, not limited at all], role-physical [1=all of the time to 5=none of the time], bodily pain [1=very severe to 6=none], general health [1=poor to 5=excellent], vitality [1=none of the time to 5=all of the time], social functioning [1=all of the time: to 5=none of the time], role emotional [1=all of the time to 5=none of the time] and mental health [1=all of the time to 5=none of the time]). Four domains comprised physical component summary (PCS) score (physical functioning, role-physical, bodily pain, general health) and remaining 4 domains comprised mental component summary (MCS) score (vitality, social functioning, role-emotional, mental health). The scores ranged from 0 to 100. Higher scores indicating better HRQL.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 50 | 104 | 106
Score on a Scale
  Physical Component Summary: Change at Week 12 | 4.84 (0.982) | 6.45 (0.721) | 5.54 (0.709)
  Mental Component Summary: Change at Week 12 | 2.09 (1.301) | 7.37 (0.949) | 6.68 (0.935)

22. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF-36), Version 2, Acute (Individual Domain Scores) at Week 12
Description: SF-36 was a generic quality-of-life instrument that had been widely used to assess HRQL of participants. Generic instruments were used in general populations to assess a wide range of domains applicable to a variety of health states, conditions, and diseases. The SF-36 consisted of 36 items that were aggregated into 8 multi-item scales (physical functioning [1=yes, limited a lot to 3=no, not limited at all], role-physical [1=all of the time to 5=none of the time], bodily pain [1=very severe to 6=none], general health [1=poor to 5=excellent], vitality [1=none of the time to 5=all of the time], social functioning [1=all of the time: to 5=none of the time], role emotional [1=all of the time to 5=none of the time] and mental health [1=all of the time to 5=none of the time]), with scores ranged from 0 to 100. Higher scores indicating better HRQL.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 50 | 104 | 106
Score on a Scale
  Physical Functioning: Change at Week 12 | 3.40 (0.901) | 5.03 (0.657) | 3.79 (0.646)
  Role-Physical: Change at Week 12 | 4.47 (1.205) | 7.39 (0.884) | 6.90 (0.874)
  Bodily Pain: Change at Week 12 | 5.55 (1.293) | 8.18 (0.941) | 7.06 (0.926)
  General Health: Change at Week 12 | 3.93 (1.203) | 7.00 (0.880) | 6.34 (0.865)
  Vitality: Change at Week 12 | 3.59 (1.381) | 8.23 (1.008) | 7.43 (0.993)
  Social Functioning: Change at Week 12 | 3.59 (1.233) | 7.43 (0.898) | 6.54 (0.884)
  Role-Emotional: Change at Week 12 | 1.27 (1.317) | 5.79 (0.958) | 5.68 (0.944)
  Mental Health: Change at Week 12 | 3.56 (1.268) | 7.90 (0.925) | 6.47 (0.911)

23. Secondary Outcome: Number of Participants Based on Inpatient Hospitalization
Description: Number of participants based on inpatient hospitalization due to all-cause hospitalization, gastrointestinal related, other illness/problem, and undergo gastrointestinal related procedures during the entire study period were reported.
Time Frame: From start of study up to follow up (Week 29)
Population: FAS consisted of all participants in the randomized set who had received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 56 | 111 | 112
Participants
  All-Cause Hospitalization | 2 | 3 | 2
  Gastrointestinal Related | 1 | 2 | 1
  Other Illness/Problem | 1 | 2 | 2
  Undergo Gastrointestinal Related Procedures | 1 | 0 | 0

24. Secondary Outcome: Median Duration of Total Inpatient Days
Description: Inpatient days were calculated as Date of discharge - Date of admission + 1. Median duration of total inpatient days during the entire study period was reported.
Time Frame: From start of study up to follow-up (Week 29)
Population: as for outcome 13
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
Number analyzed (Participants) | 2 | 3 | 2
Days | 10.5 [6 to 15] | 7.0 [6 to 11] | 2.0 [2 to 2]

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (Week 29)
Groups:
- Placebo: Participants received placebo matched to ontamalimab subcutaneous (SC) injection using a prefilled syringe (PFS) on Week 0, Week 4, and Week 8.
- Ontamalimab 25 mg: Participants received 25 milligram (mg) of ontamalimab SC injection using a PFS on Week 0, Week 4 and Week 8.
- Ontamalimab 75 mg: Participants received 75 mg of ontamalimab SC injection using PFS on Week 0, Week 4 and Week 8.
Arm/Group | Placebo | Ontamalimab 25 mg | Ontamalimab 75 mg
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/111 | 0/112
Serious Adverse Events (participants affected / at risk) | 4/56 | 5/111 | 3/112
Other Adverse Events (participants affected / at risk) | 7/56 | 5/111 | 7/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=56) | Ontamalimab 25 mg (N=111) | Ontamalimab 75 mg (N=112)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocalyx (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=56) | Ontamalimab 25 mg (N=111) | Ontamalimab 75 mg (N=112)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 2 (2) | 7 (9)
Nausea (Gastrointestinal disorders) | 4 (5) | 3 (3) | 2 (3)

LIMITATIONS AND CAVEATS:
The study was terminated as per the sponsor decision to discontinue the SHP647 (ontamalimab) clinical trial development program for inflammatory bowel diseases (IBD) early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT03259308/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT03259308/SAP_001.pdf